CLINICAL TRIAL: NCT00272584
Title: International Study of Improving Treatment for the Most Severely Ill With Schizophrenia
Brief Title: CARE Study: Improving Treatment for the Most Severely Ill With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C0-0280
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2006-05-08 (Estimated); Status verified 2006-01

CONDITIONS: Psychosis, Schizophrenia
Keywords: Psychosis, schizophrenia, schizoaffective, clozapine, risperidone
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
This is a 9 week, multicentre, randomized, double-blind, placebo-controlled trial with two parallel groups. There is also an open-label extension phase of 18 weeks. Both medications to be used in the study, clozapine and risperidone, are fully approved for the treatment of schizophrenia.

DETAILED DESCRIPTION:
Subjects may be inpatients or outpatients. All subjects will be treated throughout the study with clozapine, at a dose of 400 mg or more, unless limited by side effects. After screening, subjects will be augmented with placebo for 7 days. Any subject with a reduction in PANSS total score of 20% or greater will be discontinued from the study. Beginning on day 8, subjects will be randomized to continued augmentation of clozapine with placebo, or to augmentation with risperidone. The initial daily dose of risperidone will be 1.0 mg, increased in 1.0 mg increments to a total of 3.0 mg/day over a two week period. Subjects unable to tolerate at least one tablet of study medication will be dropped from the study. At the end of 8 weeks following randomization, at the choice of the investigator, open-label risperidone augmentation can be started.

The primary outcome measure is the PANSS total score at week 9. Subjects will be classified as responders if the improvement in PANSS total score is 20% or greater, and the proportion of responders in each group will be determined. Complementary outcome measures will be the CGI severity score, CGI improvement score, and SOFAS score. Safety and tolerance will be assessed by reports of adverse events and clinically significant changes in vital signs, weight, waist circumference, extrapyramidal side effects, metabolic and hematological measures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects treated with clozapine for the indication of poor response to other antipsychotic medications.
* Treatment with clozapine is at a stable dose for at least 12 weeks. Dose must be 400 mg/day or more, unless side effects limited increase of dose.

Exclusion Criteria:

* Subjects with significant alcohol or substance abuse in the past 3 months.
* Subjects with a previous trial of risperidone augmentation of clozapine
* Subjects who are pregnant, breast-feeding, or women of child-bearing potential not using adequate contraception
* Subjects requiring treatment with anticonvulsants.
* Subjects with known hypersensitivity or allergy to risperidone.
* Subjects with hematological or other contraindications to continued clozapine treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-06; Study Completion 2004-01

PRIMARY OUTCOMES:
For 100 subjects with incomplete response to adequate treatment with clozapine, the primary objective is to determine if risperidone augmentation of clozapine is superior to augmentation with placebo, using the outcome measure of total PANSS score

SECONDARY OUTCOMES:
Additional outcome measures will be: proportion of subjects with a 20% or greater reduction in PANSS total score, CGI severity score, CGI improvement score and SOFAS score.
To assess the safety of risperidone augmentation, severity of extrapyramidal side effects, metabolic measures, and general side effects will be studied. Hematological monitoring will be carried out.
To determine if risperidone augmentation has effects on cognition, a neuropsychological test battery will be carried out.
The predictive value of neurocognitive testing, and DNA analysis for results of risperidone augmentation will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: William Honer, MD, Principal Investigator — University of British Columbia
Locations (1):
- UBC Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Honer WG, Thornton AE, Chen EY, Chan RC, Wong JO, Bergmann A, Falkai P, Pomarol-Clotet E, McKenna PJ, Stip E, Williams R, MacEwan GW, Wasan K, Procyshyn R; Clozapine and Risperidone Enhancement (CARE) Study Group. Clozapine alone versus clozapine and risperidone with refractory schizophrenia. N Engl J Med. 2006 Feb 2;354(5):472-82. doi: 10.1056/NEJMoa053222. PMID 16452559
- [Derived] Thornton AE, Procyshyn RM, Barr AM, MacEwan GW, Honer WG. Cognition and Plasma Ratio of Clozapine to N-desmethylclozapine in Patients With Clozapine-Resistant Schizophrenia. Am J Psychiatry. 2015 Dec;172(12):1259. doi: 10.1176/appi.ajp.2015.15070899. No abstract available. PMID 26619773